CLINICAL TRIAL: NCT00985790
Title: Immunogenicity and Safety Study of a GlaxoSmithKline Biologicals' Candidate Influenza Vaccine GSK2321138A in Healthy Children
Brief Title: Immunogenicity and Safety Study of a GlaxoSmithKline Biologicals' Candidate Influenza Vaccine in Healthy Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113237
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: vaccine; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- GSK2321138A Group (Experimental): Subjects aged between 18 and 47 months received the GSK2321138A. "Primed" subjects (subjects who had received a 2-dose priming immunization with Fluarix™ vaccine in study NCT00764790 - or the GSK2321138A-Primed Group) received 1 dose of GSK2321138A vaccine at Day 0. "Unprimed" subject (subjects who had not received any 2-dose priming influenza immunization in any previous year - or the the GSK2321138A-Unprimed Group) received 2 doses of GSK2321138A vaccine at Days 0 and 28. The GSK2321138A vaccine was administered intramuscularly in the deltoid of the right arm.
  Interventions: Biological: Influenza vaccine GSK2321138A
- Fluarix Group (Active Comparator): Subjects aged between 18 and 47 months received the Fluarix™ vaccine. "Primed" subjects (subjects who had received a 2-dose priming immunization with Fluarix™ vaccine in study NCT00764790 - or the Fluarix-Primed Group) received 1 dose of Fluarix™ vaccine at Day 0. "Unprimed" subject (subjects who had not received any 2-dose priming influenza immunization in any previous year - or the the Fluarix-Unprimed Group) received 2 doses of Fluarix™ vaccine at Days 0 and 28. The Fluarix™ vaccine was administered intramuscularly in the deltoid of the right arm.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Influenza vaccine GSK2321138A — Intramuscular injection
  Arms: GSK2321138A Group
Biological: Fluarix™ — Intramuscular injection
  Arms: Fluarix Group

SUMMARY:
The purpose of the present study is to assess the immunogenicity and safety of vaccine GSK2321138A in children.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Subjects who the investigator believes that they and/or their Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject/from the LAR(s).

For unprimed subjects:

* A male or female child aged 18 to 47 months at the time of the first vaccination.
* Children who did not have influenza vaccine in a previous season.

For primed subjects from study NCT00764790:

• Children who received Fluarix™ in the 111751 study NCT00764790.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* History of hypersensitivity to any vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before and ending 28 days after each dose of vaccine(s).
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Acute disease at the time of enrolment.
* History of Guillain Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Receipt of another seasonal influenza vaccine outside of this study, during current (2009-2010) flu season.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccination Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or blood products within the 3 month preceding the first dose of study vaccine or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.

Ages: 18 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 599 (Actual)
Dates: Start 2009-10-08; Primary Completion 2010-05-21 (Actual); Study Completion 2010-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Mexico (2):
  - GSK Investigational Site, Ecatepec de Morelos, State of Mexico
  - GSK Investigational Site, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Rodriguez Weber MA, Claeys C, Aranza Doniz C, Feng Y, Innis BL, Jain VK, Peeters M. Immunogenicity and safety of inactivated quadrivalent and trivalent influenza vaccines in children 18-47 months of age. Pediatr Infect Dis J. 2014 Dec;33(12):1262-9. doi: 10.1097/INF.0000000000000463. PMID 25386965
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 113237 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113237 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113237 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113237 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113237 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113237 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 599 subjects were enrolled in the study, and assigned to either the GSK2321138A Group (298 subjects) or the Fluarix Group (301 subjects). Duration of study was of approximately 6 months for each subject.
Pre-assignment Details: For demography and safety, results are presented as per the main study groups. For some outcome measures and where relevant, subjects as in these 2 main groups are split according to their priming status at study entry.
Period: Overall Study
Arm/Group | GSK2321138A Group | Fluarix Group
Started | 298 (95 were primed and 203 were unprimed subjects.) | 301 (97 were primed and 204 were unprimed subjects.)
Completed | 291 | 293
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2321138A Group | Fluarix Group | Total
Number analyzed (Participants) | 298 | 301 | 599
Age, Continuous [Mean (Standard Deviation); unit: months] | 31.4 (8.46) | 31.6 (8.29) | 31.5 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 147 | 285
  Male | 160 | 154 | 314

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the 3 Fluarix Vaccine Strains.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. The 3 influenza strains assessed were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2) and Flu B/Brisbane/60/08 Victoria (VICT).The POST results were the primary outcome variables.
Time Frame: At Day 0 [PRE] and at 28 days post last vaccination (Day 28 or Day 56) [POST]
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK2321138A Group | Fluarix Group
Number analyzed (Participants) | 193 | 193
titers
  H1N1, PRE: number analyzed (Participants) | 189 | 192
  H1N1, PRE | 22.2 [17.2 to 28.7] | 21.6 [16.7 to 28.0]
  H1N1, POST | 173.8 [141.4 to 213.5] | 176.9 [143.3 to 218.5]
  H3N2, PRE: number analyzed (Participants) | 190 | 192
  H3N2, PRE | 18.6 [14.9 to 23.2] | 20.8 [16.5 to 26.2]
  H3N2, POST | 120.7 [101.2 to 143.9] | 130.4 [108.0 to 157.5]
  VICT, PRE: number analyzed (Participants) | 190 | 192
  VICT, PRE | 8.7 [7.3 to 10.2] | 9.0 [7.7 to 10.6]
  VICT, POST: number analyzed (Participants) | 192 | 193
  VICT, POST | 61.9 [48.7 to 78.6] | 66.6 [52.4 to 84.7]

2. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. The 4 influenza strains assessed were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the primed groups.
Time Frame: At Days 0 and 28.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- GSK2321138A-Primed Group: Subjects in this group were the primed subjects from the GSK2321138A Group, aged between 18 and 47 months, who received 1 dose of GSK2321138A vaccine at Day 0, and who had previously received a 2-dose priming immunization with Fluarix™ vaccine in study NCT00764790. The GSK2321138A vaccine was administered intramuscularly in the deltoid of the right arm.
- Fluarix-Primed Group: Subjects in this group were the primed subjects from the Fluarix Group, aged between 18 and 47 months, who received 1 dose of Fluarix™ vaccine at Day 0, and who had previously received a 2-dose priming immunization with Fluarix™ vaccine in study NCT00764790. The Fluarix™ vaccine was administered intramuscularly in the deltoid of the right arm.
Arm/Group | GSK2321138A-Primed Group | Fluarix-Primed Group
Number analyzed (Participants) | 94 | 95
titers
  H1N1. Day 0 | 40.3 [27.0 to 60.2] | 36.5 [24.3 to 54.9]
  H1N1. Day 28 | 117.0 [83.2 to 164.5] | 124.4 [89.8 to 172.4]
  H3N2, Day 0 | 22.8 [16.7 to 31.2] | 21.7 [16.0 to 29.5]
  H3N2, Day 28 | 85.2 [64.8 to 112.0] | 83.0 [63.6 to 108.2]
  VICT, Day 0 | 8.9 [7.2 to 11.0] | 9.7 [7.7 to 12.4]
  VICT, Day 28 | 38.7 [26.2 to 57.1] | 44.0 [29.6 to 65.2]
  YAMA, Day 0 | 29.3 [23.0 to 37.4] | 37.7 [29.8 to 47.8]
  YAMA, Day 28 | 243.6 [198.1 to 299.6] | 127.2 [106.1 to 152.3]

3. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. The 4 influenza strains assessed were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the unprimed groups.
Time Frame: At Days 0, 28 and Day 56
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- GSK2321138A-Unprimed Group: Subjects in this group were the unprimed subjects from the GSK2321138A Group, aged between 18 and 47 months, who received 2 doses of GSK2321138A vaccine at Days 0 and 28, and who had not received any 2-dose priming influenza immunization in any previous year. The GSK2321138A vaccine was administered intramuscularly in the deltoid of the right arm.
- Fluarix-Unprimed Group: Subjects in this group were the unprimed subjects from the Fluarix Group, aged between 18 and 47 months, who received 2 doses of Fluarix™ vaccine at Days 0 and 28, and who had not received any 2-dose priming influenza immunization in any previous year. The Fluarix™ vaccine was administered intramuscularly in the deltoid of the right arm.
Arm/Group | GSK2321138A-Unprimed Group | Fluarix-Unprimed Group
Number analyzed (Participants) | 192 | 198
titers
  H1N1, Day 0: number analyzed (Participants) | 190 | 198
  H1N1, Day 0 | 14.7 [11.8 to 18.4] | 12.8 [10.5 to 15.7]
  H1N1, Day 28: number analyzed (Participants) | 97 | 101
  H1N1, Day 28 | 173.1 [113.1 to 264.8] | 161.6 [103.9 to 251.4]
  H1N1, Day 56: number analyzed (Participants) | 99 | 98
  H1N1, Day 56 | 253.1 [203.4 to 314.8] | 249.0 [192.5 to 321.9]
  H3N2, Day 0: number analyzed (Participants) | 192 | 197
  H3N2, Day 0 | 17.7 [14.1 to 22.1] | 17.9 [14.1 to 22.6]
  H3N2, Day 28: number analyzed (Participants) | 96 | 101
  H3N2, Day 28 | 99.3 [64.8 to 152.2] | 84.2 [54.1 to 131.2]
  H3N2, Day 56: number analyzed (Participants) | 99 | 98
  H3N2, Day 56 | 168.1 [136.6 to 206.7] | 202.1 [158.6 to 257.5]
  VICT, Day 0: number analyzed (Participants) | 190 | 198
  VICT, Day 0 | 7.8 [6.7 to 9.2] | 8.7 [7.5 to 10.3]
  VICT, Day 28: number analyzed (Participants) | 95 | 101
  VICT, Day 28 | 26.5 [17.7 to 39.7] | 34.6 [22.4 to 53.6]
  VICT, Day 56: number analyzed (Participants) | 98 | 98
  VICT, Day 56 | 97.2 [74.9 to 126.1] | 99.6 [76.7 to 129.4]
  YAMA, Day 0: number analyzed (Participants) | 188 | 198
  YAMA, Day 0 | 9.1 [7.7 to 10.7] | 9.9 [8.4 to 11.8]
  YAMA, Day 28: number analyzed (Participants) | 97 | 102
  YAMA, Day 28 | 97.0 [64.7 to 145.4] | 30.0 [21.3 to 42.1]
  YAMA, Day 56: number analyzed (Participants) | 99 | 98
  YAMA, Day 56 | 311.1 [255.4 to 379.1] | 42.2 [30.6 to 58.1]

4. Secondary Outcome: Number of Seropositive Subjects Against 4 Strains of Influenza Disease.
Description: A seropositive subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:10. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the primed groups.
Time Frame: At Days 0 and 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A-Primed Group | Fluarix-Primed Group
Number analyzed (Participants) | 94 | 95
Participants
  H1N1, Day 0 | 58 | 54
  H1N1, Day 28 | 83 | 87
  H3N2, Day 0 | 60 | 59
  H3N2, Day 28 | 88 | 87
  VICT, Day 0 | 26 | 28
  VICT, Day 28 | 62 | 66
  YAMA, Day 0 | 73 | 80
  YAMA, Day 28 | 93 | 94

5. Secondary Outcome: Number of Seropositive Subjects Against 4 Strains of Influenza Disease.
Description: A seropositive subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:10. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the unprimed groups.
Time Frame: At Days 0, 28 and 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A-Unprimed Group | Fluarix-Unprimed Group
Number analyzed (Participants) | 192 | 198
Participants
  H1N1, Day 0: number analyzed (Participants) | 190 | 198
  H1N1, Day 0 | 75 | 71
  H1N1, Day 28: number analyzed (Participants) | 97 | 101
  H1N1, Day 28 | 83 | 84
  H1N1, Day 56: number analyzed (Participants) | 99 | 98
  H1N1, Day 56 | 99 | 96
  H3N2, Day 0: number analyzed (Participants) | 192 | 197
  H3N2, Day 0 | 85 | 82
  H3N2, Day 28: number analyzed (Participants) | 96 | 101
  H3N2, Day 28 | 74 | 78
  H3N2, Day 56: number analyzed (Participants) | 99 | 98
  H3N2, Day 56 | 99 | 98
  VICT, Day 0: number analyzed (Participants) | 190 | 198
  VICT, Day 0 | 30 | 42
  VICT, Day 28: number analyzed (Participants) | 95 | 101
  VICT, Day 28 | 51 | 61
  VICT, Day 56: number analyzed (Participants) | 98 | 98
  VICT, Day 56 | 96 | 94
  YAMA, Day 0: number analyzed (Participants) | 188 | 198
  YAMA, Day 0 | 45 | 57
  YAMA, Day 28: number analyzed (Participants) | 97 | 102
  YAMA, Day 28 | 75 | 57
  YAMA, Day 56: number analyzed (Participants) | 99 | 98
  YAMA, Day 56 | 98 | 70

6. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the primed groups.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A-Primed Group | Fluarix-Primed Group
Number analyzed (Participants) | 94 | 95
Participants
  H1N1, Day 28 | 30 | 39
  H3N2, Day 28 | 48 | 46
  VICT, Day 28 | 46 | 42
  YAMA, Day 28 | 82 | 40

7. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the unprimed groups.
Time Frame: At Days 28 and 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A-Unprimed Group | Fluarix-Unprimed Group
Number analyzed (Participants) | 96 | 101
Participants
  H1N1, Day 28: number analyzed (Participants) | 95 | 101
  H1N1, Day 28 | 63 | 74
  H1N1, Day 56: number analyzed (Participants) | 95 | 97
  H1N1, Day 56 | 81 | 89
  H3N2, Day 28: number analyzed (Participants) | 96 | 100
  H3N2, Day 28 | 55 | 54
  H3N2, Day 56: number analyzed (Participants) | 96 | 97
  H3N2, Day 56 | 79 | 75
  VICT, Day 28: number analyzed (Participants) | 94 | 101
  VICT, Day 28 | 34 | 40
  VICT, Day 56: number analyzed (Participants) | 95 | 97
  VICT, Day 56 | 77 | 85
  YAMA, Day 28: number analyzed (Participants) | 93 | 101
  YAMA, Day 28 | 59 | 40
  YAMA, Day 56: number analyzed (Participants) | 95 | 97
  YAMA, Day 56 | 90 | 42

8. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the primed groups.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2321138A-Primed Group | Fluarix-Primed Group
Number analyzed (Participants) | 94 | 95
fold change
  H1N1, Day 28 | 2.9 [2.3 to 3.6] | 3.4 [2.7 to 4.2]
  H3N2, Day 28 | 3.7 [3.1 to 4.5] | 3.8 [3.1 to 4.7]
  VICT, Day 28 | 4.4 [3.3 to 5.8] | 4.5 [3.4 to 6.0]
  YAMA, Day 28 | 8.3 [6.8 to 10.1] | 3.4 [2.8 to 4.0]

9. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the unprimed groups.
Time Frame: At Days 28 and 56
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | GSK2321138A-Unprimed Group | Fluarix-Unprimed Group
Number analyzed (Participants) | 96 | 101
fold change
  H1N1, Day 28: number analyzed (Participants) | 95 | 101
  H1N1, Day 28 | 9.9 [7.0 to 14.1] | 12.7 [9.1 to 17.7]
  H1N1, Day 56: number analyzed (Participants) | 95 | 97
  H1N1, Day 56 | 19.8 [15.4 to 25.6] | 19.2 [15.2 to 24.2]
  H3N2, Day 28: number analyzed (Participants) | 96 | 100
  H3N2, Day 28 | 4.9 [3.7 to 6.3] | 5.1 [3.9 to 6.7]
  H3N2, Day 56: number analyzed (Participants) | 96 | 97
  H3N2, Day 56 | 11.1 [9.0 to 13.7] | 10.3 [8.3 to 12.9]
  VICT, Day 28: number analyzed (Participants) | 94 | 101
  VICT, Day 28 | 3.6 [2.7 to 5.0] | 3.8 [2.9 to 5.0]
  VICT, Day 56: number analyzed (Participants) | 95 | 97
  VICT, Day 56 | 11.3 [9.4 to 13.6] | 12.1 [9.8 to 14.8]
  YAMA, Day 28: number analyzed (Participants) | 93 | 101
  YAMA, Day 28 | 9.9 [6.9 to 14.0] | 3.4 [2.5 to 4.5]
  YAMA, Day 56: number analyzed (Participants) | 95 | 97
  YAMA, Day 56 | 35.1 [27.6 to 44.6] | 3.7 [2.9 to 4.8]

10. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the primed groups.
Time Frame: At Days 0 and 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A-Primed Group | Fluarix-Primed Group
Number analyzed (Participants) | 94 | 95
Participants
  H1N1, Day 0 | 48 | 45
  H1N1, Day 28 | 73 | 78
  H3N2, Day 0 | 39 | 36
  H3N2, Day 28 | 75 | 80
  VICT, Day 0 | 16 | 20
  VICT, Day 28 | 50 | 52
  YAMA, Day 0 | 56 | 62
  YAMA, Day 28 | 91 | 90

11. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The 4 assessed influenza strains were the FLU A/Brisbane/59/07 (H1N1), Flu A/Uruguay/716/07 (H3N2), Flu B/Brisbane/60/08 Victoria (VICT) and Flu B/Brisbane/3/07 Yamagata (YAMA). This outcome only covers the results for the unprimed groups.
Time Frame: At Days 0, 28 and 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A-Unprimed Group | Fluarix-Unprimed Group
Number analyzed (Participants) | 192 | 198
Participants
  H1N1, Day 0: number analyzed (Participants) | 190 | 198
  H1N1, Day 0 | 58 | 54
  H1N1, Day 28: number analyzed (Participants) | 97 | 101
  H1N1, Day 28 | 76 | 78
  H1N1, Day 56: number analyzed (Participants) | 99 | 98
  H1N1, Day 56 | 95 | 94
  H3N2, Day 0: number analyzed (Participants) | 192 | 197
  H3N2, Day 0 | 74 | 70
  H3N2, Day 28: number analyzed (Participants) | 96 | 101
  H3N2, Day 28 | 64 | 61
  H3N2, Day 56: number analyzed (Participants) | 99 | 98
  H3N2, Day 56 | 96 | 94
  VICT, Day 0: number analyzed (Participants) | 190 | 198
  VICT, Day 0 | 25 | 35
  VICT, Day 28: number analyzed (Participants) | 95 | 101
  VICT, Day 28 | 36 | 41
  VICT, Day 56: number analyzed (Participants) | 98 | 98
  VICT, Day 56 | 84 | 88
  YAMA, Day 0: number analyzed (Participants) | 188 | 198
  YAMA, Day 0 | 37 | 40
  YAMA, Day 28: number analyzed (Participants) | 97 | 102
  YAMA, Day 28 | 67 | 53
  YAMA, Day 56: number analyzed (Participants) | 99 | 98
  YAMA, Day 56 | 98 | 59

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling at the injection site. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day follow-up period (Days 0 to 6) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with the symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group
Number analyzed (Participants) | 293 | 298
Participants
  Any Pain | 125 | 116
  Grade 3 Pain | 4 | 1
  Any Redness | 31 | 34
  Redness >50 mm | 0 | 0
  Any Swelling | 27 | 24
  Swelling >50 mm | 0 | 0

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature (defined as axillary temperature equal to or above 37.5 degrees Celsius). For other symptoms: Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms assessed by the investigator as related to vaccination. Grade 3 drowsiness = prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 irritability= crying that could not be comforted/prevented normal activity. Grade 3 temperature: ≥ 39.0°C.
Time Frame: During the 7-day follow-up period (Days 0 to 6) after any vaccination
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group
Number analyzed (Participants) | 293 | 298
Participants
  Any Drowsiness | 70 | 62
  Grade 3 Drowsiness | 2 | 0
  Related Drowsiness | 64 | 57
  Any Irritability | 90 | 87
  Grade 3 Irritability | 4 | 2
  Related Irritability | 83 | 78
  Any Loss of appetite | 89 | 86
  Grade 3 Loss of appetite | 4 | 3
  Related Loss of appetite | 79 | 68
  Temperature ≥ 37.5°C | 74 | 79
  Temperature > 39.0°C | 3 | 3
  Related Temperature | 63 | 62

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to vaccination.
Time Frame: During the 28-day follow-up period (Days 0 to 27) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group
Number analyzed (Participants) | 298 | 301
Participants
  Subjects with any AE(s) | 116 | 118
  Subjects with Grade 3 AE(s) | 10 | 12
  Subjects with related AE(s) | 7 | 9

15. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Any was defined as occurrence of any symptom regardless of intensity grade and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 to Day 180 (study conclusion)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2321138A Group | Fluarix Group
Number analyzed (Participants) | 298 | 301
Participants
  Subjects with any SAE(s) | 0 | 2
  Subjects with related SAE(s) | 0 | 0

16. Secondary Outcome: Number of Subjects With Any Adverse Events of Specific Interest (AESIs).
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 to Day 180 (study conclusion)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2321138A Group: Subjects aged between 18 and 47 months received the GSK2321138A. "Primed" subjects (subjects who had received a 2-dose priming immunization with Fluarix™ vaccine in study NCT00764790 - or the GSK2321138A-Primed Group) received 1 dose of GSK2321138A vaccine at Day 0. "Unprimed" subject (subjects who had not received any 2-dose priming influenza immunization in any previous year - or the GSK2321138A-Unprimed Group) received 2 doses of GSK2321138A vaccine at Days 0 and 28. The GSK2321138A vaccine was administered intramuscularly in the deltoid of the right arm.
Arm/Group | GSK2321138A Group | Fluarix Group
Number analyzed (Participants) | 298 | 301
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (Day 0 - Day 180); Unsolicited AE(s): during the 28-day follow-up period (Days 0 to 27) after any vaccination; Solicited local and general symptoms: during the 7-day (Days 0-6) follow-up period after any vaccination.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed. No related SAEs were reported.
Arm/Group | GSK2321138A Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 0/298 | 2/301
Other Adverse Events (participants affected / at risk) | 230/298 | 221/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2321138A Group (N=298) | Fluarix Group (N=301)
Bronchopneumonia (Infections and infestations) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2321138A Group (N=298) | Fluarix Group (N=301)
Nasopharyngitis (Infections and infestations) | 72 | 69
Pharyngitis (Infections and infestations) | 20 | 21
Drowsiness (General disorders) | 70/293 | 62/298
Irritability (General disorders) | 90/293 | 87/298
Loss of appetite (General disorders) | 89/293 | 86/298
Temperature (General disorders) | 74/293 | 79/298
Pain (General disorders) | 125/293 | 116/298
Redness (General disorders) | 31/293 | 34/298
Swelling (General disorders) | 27/293 | 24/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.